CLINICAL TRIAL: NCT01304875
Title: Pulmonary Disease and Exercise Tolerance in Boys With Fabry Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Rare Diseases Clinical Research Network (Network); National Center for Advancing Translational Sciences (NCATS) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Genzyme, a Sanofi Company (Industry)
Responsible Party: Principal Investigator, William Wilcox, Professor of Pediatrics, Cedars-Sinai Medical Center
Other Study IDs: CSMC17883; U54NS065768 (NIH)
Record Dates: First submitted 2011-02-25; First posted 2011-02-28 (Estimated); Last update posted 2013-06-27 (Estimated); Status verified 2013-06

CONDITIONS: Fabry Disease
Keywords: Fabry disease; alpha-galactosidase deficiency; exercise; pulmonary
MeSH Terms: conditions — Fabry Disease; Motor Activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
When to start children with Fabry disease on therapy is controversial because of its expense and inconvenience. Many Fabry children complain of exercise intolerance. In adults, the investigators have found decreased lung function and ability to exercise on a treadmill. Whether or not lung function and exercise capacity is abnormal in children is unknown. While lung function and exercise tests are commonly part of routine evaluations for adults with Fabry, they are not yet for children.

The objective of the proposed study is to more accurately define the lung and exercise abnormalities in a group of 20 boys from 8-18 years of age with Fabry disease who have not been treated with enzyme replacement therapy (Fabrazyme).

DETAILED DESCRIPTION:
Fabry disease is due to an alteration in the genetic material (DNA) that causes a deficiency of the alpha-galactosidase A enzyme. This enzyme aids in the breakdown and elimination of certain types of fatty substances called glycolipids. These glycolipids are normally present within the body in most cells. When alpha-galactosidase A is lacking, these glycolipids build up in various tissues such as the eye, liver, kidney, skin, muscle, heart, and blood vessels. The build up of glycolipid levels in these tissues, particularly globotriaosylceramide (GL-3), is thought to cause the clinical symptoms that are associated with Fabry disease. Fabry disease causes chronic kidney damage leading to a need for dialysis or kidney transplantation, chronic heart damage leading to abnormal heart rhythms and heart attacks and strokes at an early age, nervous system damage leading to chronic pain, and a premature death. Because the gene for Fabry is on the X chromosome (men have only one X chromosome while women have two), most patients with symptoms of Fabry are men but many women have symptoms that may be as severe as men. There is currently a FDA approved treatment available that treats many of the symptoms of Fabry, but it involves intravenous infusions every other week and is very expensive.

When to start children on therapy is controversial because of its expense and inconvenience. Children with significant pain or gastrointestinal problems are started on therapy immediately, otherwise not until they are at least teenagers. Increasing evidence suggests that even without overt symptoms, significant, irreversible damage may be occurring in childhood. However, determining whether such damage is present or not requires biopsies. There are no simple measures of disease severity.

Many Fabry children complain of exercise intolerance. In adults, the investigators have found decreased lung function and ability to exercise on a treadmill. Whether or not lung function and exercise capacity is abnormal in children is unknown. While lung function and exercise tests are commonly part of routine evaluations for adults with Fabry, they are not yet for children.

The objective of the proposed study is to more accurately define the lung and exercise abnormalities in a group of 20 boys from 8-18 years of age with Fabry disease who have not been treated with enzyme replacement therapy (Fabrazyme). This will be done by several breathing tests and exercising on a treadmill. If the breathing tests are abnormal, then testing would serve as an easy way to evaluate children and help decide when therapy should be started and monitor the effectiveness of therapy.

Each person that consents to participate in the study will be required to commit to a single study visit that will last approximately 4 hours at Cedars-Sinai Medical Center. The participant will be expected to wear loose fit clothing and comfortable athletic footwear.

As part of the research, participants will be asked to participate in the following tests:

1. A pulmonary function test
2. Exercise test. Results will be forwarded to each participant's primary care physician.

All subjects must have previously been enrolled in the Fabry Registry and have the recommended standard of care assessments in order to be eligible for this pilot study.

ELIGIBILITY:
Inclusion Criteria:

* Fabry disease
* Male
* Between 8-18 years of age
* Enrolled in Fabry registry and have standard assessments

Exclusion Criteria:

* Enzyme replacement therapy or an experimental therapy
* Inability to perform the tests
* Other, serious medical conditions that would impact the tests

Ages: 8 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Boys between ages 8 and 18 years of age with Fabry disease not receiving enzyme replacement therapy or an experimental therapy.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2010-04

PRIMARY OUTCOMES:
Measurement of pulmonary function | upon enrollment
  Research subjects' pulmonary function will be determined by FEF25-75, VO2 max, and treadmill studies.

SECONDARY OUTCOMES:
Measurement of diastolic blood pressure | upon enrollment
  The maximum decrease in diastolic blood pressure with exercise will be compared to baseline diastolic blood pressure.

CONTACTS AND LOCATIONS:
Overall Officials: William R Wilcox, MD, PhD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States